CLINICAL TRIAL: NCT04260165
Title: A Double-blinded Randomized Controlled Multicenter Trial Comparing Proximal ROw carpectOmy and Four-corner Fusion (PROOF) for Osteoarthritis of the Wrist
Brief Title: Proximal Row Carpectomy vs Four-corner Fusion for Osteoarthritis of the Wrist
Acronym: PROOF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Töölö Hospital (Other)
Collaborators: Tampere University Hospital (Other); Turku University Hospital (Other Government); Jyväskylä Central Hospital (Other); Kymenlaakso Central Hospital Kotka Finland (Other)
Responsible Party: Principal Investigator, Samuli Aspinen, Principal investigator, Töölö Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUS/3487/2019
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Wrist Osteoarthritis; Scapholunate Advanced Collapse
Keywords: Wrist Osteoarthritis; Scapholunate Advanced Collapse; Scaphoid Non-union Advanced Collapse; Wrist arthrodesis; Proximal Row Carpectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proximal Row Carpectomy (Experimental)
  Interventions: Procedure: Proximal Row Carpectomy
- Four-corner fusion (Active Comparator)
  Interventions: Procedure: Four-corner fusion

INTERVENTIONS:
Procedure: Proximal Row Carpectomy — Excision of the proximal carpal row - the scaphoid, lunate and triquetrum
  Arms: Proximal Row Carpectomy
Procedure: Four-corner fusion — Scaphoid excision and four-corner fusion with cannulated headless compression screws/dorsal plate
  Arms: Four-corner fusion

SUMMARY:
Study purpose is to compare the outcome after proximal row carpectomy (PRC) vs four-corner fusion (FCA) for SLAC/SNAC II-III type osteoarthritis (OA) in a double-blinded randomized controlled study setting.

Patients with radiologically and clinically confirmed OA are randomized (1:1 computer generated sequence with random block size) to two parallel groups and will undergo either PRC or FCA. The study will be patient and assessor blinded.

Baseline data is collected preoperatively and is followed by a follow-up visits at 2 and 6 weeks, 3, 6, 12 months, and 5, 10 years after the intervention. Unveiling of the allocation is at 12 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* SLAC/SNAC II-III
* Age 18 - 75
* Symptom duration > 3 months
* American Society of Anaesthesiologists physical status (ASA) I-II

Exclusion Criteria:

* Patient eligible for SL reconstruction or scaphoid
* Ulnocarpal/pancarpal arthritis
* Lunate fossa, proximal lunate arthrosis or both
* Age <18 or >75 years
* Rheumatoid arthritis
* Heavy smoking (> 20 cigarettes per day)
* Condition or medication affecting bony healing (eg diabetes mellitus with poor glycemic control, malnutrition, use of per oral corticosteroids)
* Alcohol or drug abuse
* Neurological condition affecting upper limb function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Rated Wrist Evaluation | 12 months
  The PRWE comprises 15 questions to measure wrist pain and disability in daily activities. In PRWE patients rate wrist pain and disability from 0 to 10 and it consists two subscales: Pain and Function (0=best possible outcome, 10=worst possible outcome)

SECONDARY OUTCOMES:
Quick-Disabilities of the Arm, Shoulder and Hand | 12 months
  The QuickDASH is self-reported questionnaire and shortened version of DASH outcome measure to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb in 11 dimensions in 1-5 scale (1=best possible outcome, 5=worst possible outcome)
Pain (Visual Analogue Scale) | 12 months
  The VAS is derived by health care professional question of pain in scale 0 to 10 (0=no pain, 10=worst possible pain)
Global improvement | 12 months
  Global rating to treatment effect will be evaluated by question: "How would you rate the function of your hand compared to the situation before the treatment?". The options are in 5-step Likert scale from (-2) Much worse to (+2) Much better
Grip strength | 12 months
  Grip strength is measured with a dynamometer in kg as the mean of three measurements. It will be numbered in kg and percentage of the unaffected side
Wrist range of motion (ROM) | 12 months
  Wrist ROM is measured on both wrists with a handheld goniometer in degrees.
Complications | 12 months
  Incidence of complications (i.e. non-union, fracture, reoperation, infection, hematoma, iatrogenic tendon/nerve/arterial injury, complex regional pain syndrome) is recorded and compared between study groups.
Patient-rated Quality of Life (EQ-5D) | 12 months
Cost-effectiveness | 12 months
  Quality-adjusted life years/months measured as a change in EQ-5D

CONTACTS AND LOCATIONS:
Locations (5):
- Finland (5):
  - Töölö Hospital (Helsinki University Hospital), Helsinki
  - Central Hospital of Central Finland, Jyväskylä
  - Kymenlaakso Central Hospital, Kotka
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alanen M, Stjernberg-Salmela S, Waris E, Karjalainen T, Miettunen J, Ryhanen J, Aspinen S. Proximal ROw carpectOmy versus four-corner Fusion (PROOF-trial) for osteoarthritis of the wrist: study protocol for multi-institutional double-blinded randomized controlled trial. Trials. 2023 Aug 7;24(1):499. doi: 10.1186/s13063-023-07544-1. PMID 37550711